CLINICAL TRIAL: NCT05650398
Title: Changes in Tactile Perception in People With Segmental Exclusion Syndrome
Status: Completed | Type: Observational
Sponsor: Union de Gestion des Etablissements des Caisses d'Assurance Maladie - Nord Est (Other)
Responsible Party: Sponsor
Other Study IDs: IRR-CLP-2022-9
Record Dates: First submitted 2022-12-05; First posted 2022-12-14 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Upper Limb Exclusion Syndrom

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with exclusion: Evaluation of the tactile sensitivity of the excluded finger using different tests: Static and dynamic two-points discrimination tests, the Semmes-Weinstein monofilament test, grating orientation task and the bar test inspired by the study of Louw et al.
  Realization of the same tests on the controllateral healthy finger.
- Control: Evaluation of the tactile sensitivity of the finger using different tests: Static and dynamic two-points discrimination tests, the Semmes-Weinstein monofilament test, grating orientation task and the bar test inspired by the study of Louw et al.
  Realization of the same tests on the controllateral finger.

SUMMARY:
Segmental exclusion syndrome is characterised by the non-use or under-use of a limb segment, most oftenly reported in the distal part, following an injury, without affecting the central nervous system. This syndrome has an important negative impact on the daily life of affected subjects; however, it remains poorly studied, particularly in terms of pathophysiology, and its management is still not specific. Currently, the main pathophysiological hypothesis is an alteration of the afferences related to a dysfunction of the sensorimotor loop. An hypothesis is that this dysfunction could concern the level of tactile perception and that the damage to the distal light touch receptors could play a role in the pathophysiology. The protocol is based on the performance of tests that explore different aspects of light touch: passive, active, dynamic and static sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* No history of upper limb involvement
* Confirmed diagnosis of segmental exclusion > 3 months after injury (2 items assigned to 400 points)
* Able to understand simple orders

Exclusion Criteria:

* Central neurological involvement after the initial or pre-existing injury
* Truncal nerve damage
* Presence of psychiatric pathology
* Communication and/or comprehension disorders
* Presence of other pathology that may lead to sensory disorders (complicated diabetes, ductal syndrome, ...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adults with a segmental exclusion of a finger more than 3 months after the initial injury. In order to study sensitivity disorders related to the exclusion, we decided to include only people who had no pathology that could have an impact on sensitivity and who had no truncal nerve damage at the time of the initial injury.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Difference in passive sensitivity discrimination orientation threshold between each hand in static condition. | once during the one-day evaluation session
  Difference in thresholds of sensitive discrimination between the two hands in the Grating Orientation Task (mm)
Difference in passive sensitivity discrimination threshold between each hand in static condition. | once during the one-day evaluation session
  Difference in thresholds of sensitive discrimination between the two hands in the Static Two Points discrimination test (mm)
Difference in passive sensitivity discrimination of pressure threshold between each hand in static condition. | once during the one-day evaluation session
  Difference in thresholds of sensitive discrimination between the two hands in the monofilament test (Newton)
Difference in passive sensitivity discrimination threshold between each hand in dynamic condition. | once during the one-day evaluation session
  Difference in thresholds of sensitive discrimination between the two hands in Moving Two-Points Discrimination Test (mm)

SECONDARY OUTCOMES:
Difference in active sensitivity discrimination threshold between each hand in dynamic condition. | During the evaluation session
  Percentage of correct answers to the bar test in both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Régional de Médecine Physique et de Réadaptation, Nancy, France